CLINICAL TRIAL: NCT01783613
Title: Study of the Eficacy of Long-term Suplementation With Docosahexaenoic Acid on Pulmonary, Sistemic and Intestinal Inflammation in Patients With Cystic Fibrosis
Brief Title: Eficacy of Long-term Suplementation With Docosahexaenoic Acid in Patients With Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Docosahexaenoic acid
Record Dates: First submitted 2013-01-31; First posted 2013-02-05 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2015-01

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Docosahexaenoic acid administration (Experimental): 50 patients will receive docosahexaenoic acid
  Interventions: Dietary Supplement: Docosahexaenoic acid administration: 50 mg/kg/day during 12 months
- placebo (Placebo Comparator): 50 patients will receive placebo
  Interventions: Dietary Supplement: Placebo: 50 mg/kg/day during 12 months

INTERVENTIONS:
Dietary Supplement: Docosahexaenoic acid administration: 50 mg/kg/day during 12 months
  Arms: Docosahexaenoic acid administration
Dietary Supplement: Placebo: 50 mg/kg/day during 12 months
  Arms: placebo

SUMMARY:
Cystic Fibrosis (CF) is a congenital disease secondary to the abnormal function of CFTR. Patients with CF have an alteration of essential fatty acids, Arachidonic Acid (AA) is increased and Docosahexanoic Acid (DHA) is decrease and the ratio ω-6/ ω-3 is elevated, all these alterations stimulated a chronic and bad regulated state of inflammation. For this porpoise, a fase IV trial, multicentric, controlled, double blind, placebo and parallel in patients elder than two months old and randomized to received every day a dietetically supplement with DHA or placebo, will be done during 12 months. The trial has as a principal objective to proved if this long term supplementation could decrease in contrast with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed of cystic fibrosis over than 2 months age
* Tolerance clinical supplementation with DHA
* Clinical situation stable

Exclusion Criteria:

* Changes in the routine treatment in the 2 weeks prior to baseline
* Admission to hospital or administration of oral or intravenous antibiotics within 2 weeks before inclusion

Ages: 2 Months to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2011-10; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
To study whether long-term administration of DHA (12 months), at doses of 50 mg/ kg/day in patients over 2 months age diagnosed of CF decreases inflammation compared with placebo | 12 months

CONTACTS AND LOCATIONS:
Locations (5):
- Spain (5):
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Ramón y Cajal Hospital, Madrid
  - Hospital 12 de Octubre, Madrid
  - Hospital Universitario La Princesa, Madrid
  - Hospital Universitari i Politecnic La FE, Valencia

REFERENCES:
- [Derived] Lopez-Neyra A, Suarez L, Munoz M, de Blas A, Ruiz de Valbuena M, Garriga M, Calvo J, Ribes C, Giron Moreno R, Maiz L, Gonzalez D, Bousono C, Manzanares J, Pastor O, Martinez-Botas J, Del Campo R, Canton R, Roy G, Menacho M, Arroyo D, Zamora J, Soriano JB, Lamas A. Long-term docosahexaenoic acid (DHA) supplementation in cystic fibrosis patients: a randomized, multi-center, double-blind, placebo-controlled trial. Prostaglandins Leukot Essent Fatty Acids. 2020 Nov;162:102186. doi: 10.1016/j.plefa.2020.102186. Epub 2020 Oct 1. PMID 33038833